CLINICAL TRIAL: NCT02046993
Title: Effect of Smart Phone Based Telemonitoring on Blood Pressure Among Hypertensive Patients in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Lorna Ventura Ng, Senior Medical Officer, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KW/EX-13-026(60-09); HKCFPRFG2013 (Other: HKCFP Research Fellowship Grant 2013)
Record Dates: First submitted 2014-01-25; First posted 2014-01-28 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension; Blood Pressure
Keywords: Hypertension; self blood pressure monitoring; smartphone based telemonitoring; primary care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smart phone based telemonitoring of HBP (Experimental): 1. . Patients do HBP monitoring
  2. . record their BP readings into the smart phone with downloaded application.
  Interventions: Behavioral: Smart phone telemonitoring HBP + enhanced usual care; Behavioral: Enhanced usual care
- Enhanced usual care (Active Comparator): 1. . Patients to do HBP measurement
  2. . Record BP readings in their diary
  Interventions: Behavioral: Smart phone telemonitoring HBP + enhanced usual care; Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Smart phone telemonitoring HBP + enhanced usual care — Smart phone telemonitoring home Blood pressure (HBP) Patients input their HBP readings to their smart phone which is sent to the data center regulary
Behavioral: Enhanced usual care — Encouraged to do HBP measurement and record BP readings in paper diary

SUMMARY:
To test the hypothesis that hypertensive patients who participate in smart phone based telemonitoring of BP will conduct more home blood pressure monitoring, better self management behavior and greater reduction in blood pressure and better self management behaviour from baseline to 6 months follow up than those patients receiving enhanced usual care.

DETAILED DESCRIPTION:
A prospective, block randomized controlled 6 months study comparing the blood pressure control of hypertensive patients who participate in enhanced usual care plus smart phone based telemonitoring (TM) of Blood Pressure (BP) to hypertensive patients receiving enhanced usual care (UC) alone in primary care setting.A previous local study done by Fung et al showed a mean diastolic BP reduction of 3.84 mmHg using manual recording of HBPM after structured program. On the basis of the expectation of least 5 mmHg difference with a power of 90% at a significance of level of 5% assuming a standard deviation of 10 mmHg and accounting for 20% attrition rate, a sample size of 206 was needed. Following the inclusion and exclusion criteria, subjects will be recruited on voluntary basis for this study. Having obtained informed consent, all subjects will be required to attend a structured home blood pressure monitoring education program based on Fung et al study and all are required to pass the self-BP measurement competency test before randomisation.[1] All participating subjects will be allocated using block randomization into the intervention group (TM) or control group (UC). Research assistants doing the assessments at baseline, 3 months and 6 months post intervention will be partially blinded to the groupings.At baseline and follow-up visits, research assistants who are blinded to allocation outcomes will measure clinic blood pressure after 15 minutes rest with validated electronic automated sphygmomanometer and conduct the self-efficacy for managing chronic disease scale ( 6-item scale). Four blood pressure readings taken at 1 minute interval will done for each subject and the mean of the 2nd and 3rd readings would be used for the outcome measures at baseline, 3 months and 6 months. For intervention group, patients will be assisted to download a mobile application tool (apps), specifically developed for use in telerecording of readings from home self BP measurement. For the control group, patients will be encouraged on self BP monitoring and keep the BP diary. The research assistants are not blinded in the collection of the mean systolic and diastolic home blood pressure readings readings based on the subjects' paper records for control group or mean systolic and diastolic BP readings sent to the data center at baseline, 3 months and 6 months. Regular home BP monitoring is defined as taking at least 3 or more BP readings per week and documented manually in their paper record or sent electronically through mobile apps to the data center.

Comparisons between these two groups in terms of compliance to home BP measurement and readings,proportion of patients doing home BP monitoring,self-efficacy outcomes and improvement in clinic BP readings at 3 months and 6 months post-intervention will be assessed using statistical analysis.Data analyses were conducted using the Statistical package for the Social Sciences (SPSS) version 16.0. Descriptive statistics, including frequency and percentage for categorical variables and mean and standard deviation for continuous variable, were used to describe the demographic characteristics and summarize baseline characteristics of the variables. Independent T-test was used to examine the differences of outcome variables between TM and UC group. A p-value of 0.05 was used as the level of statistical significance.

The principal investigator and sub-investigator will do regular monitoring, conduct regular meetings with research team to ensure quality assurance in patient recruitment, data collection, data management, data analysis, reporting for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. All hypertensive patients aged 30 or above and using smart phone
2. Agrees to participate in this pilot study
3. required to attend structured HBPM education program and assessed competent in self BP measurement

Exclusion Criteria:

1. Patients could not use the smart phone independently, such as mentally or physically incapacitated.
2. Patients are not competent in verbal or written communication.

   -

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kwong Wah Hospital General Out-Patient and Family Medicine Department, Hong Kong, Kowloon, Hong Kong, Hong Kong

REFERENCES:
- [Background] Fung CS, Wong WC, Wong CK, Lee A, Lam CL. Home blood pressure monitoring--a trial on the effect of a structured education program. Aust Fam Physician. 2013 Apr;42(4):233-7. PMID 23550251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment of eligible subjects from January to December 2014 at a primary care clinic in Hong Kong
Groups:
- Smart Phone Based Telemonitoring of HBP + Enhanced Usual Care: Smart phone based telemonitoring home blood pressure (HBP)
  1. . Patients do HBP monitoring
  2. . record their BP readings into the smart phone with downloaded application.
  Smart phone telemonitoring HBP: Smart phone telemonitoring home Blood pressure (HBP) Patients to do home BP measurement and input into their smart phone which is sent to the central server fortnightly
- Hypertensive Patients on Enahnced Usual Care: Hypertensive patients on usual care
  1. . Patients to do HBP measurement
  2. . Record BP readings in their diary
  Hypertensive patient on usual care: Patient do home BP monitoring Record the Home BP monitoring in their diary
Period: Overall Study
Arm/Group | Smart Phone Based Telemonitoring of HBP + Enhanced Usual Care | Hypertensive Patients on Enahnced Usual Care
Started | 105 | 105
3rd Month | 104 | 97
6th Month | 102 | 94
Completed | 102 | 94
Not Completed | 3 | 11
Not completed — Withdrawal by Subject | 2 | 10
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Smart Phone Based Telemonitoring of HBP: Smart phone based telemonitoring home blood pressure (HBP)
  1. . Patients do HBP monitoring
  2. . record their BP readings into the smart phone with downloaded application.
  Smart phone telemonitoring HBP: Smart phone telemonitoring home Blood pressure (HBP) Patients to do home BP measurement and input into their smart phone which is sent to the central server fortnightly
- Hypertensive Patients on Usual Care: Hypertensive patients on usual care
  1. . Patients to do HBP measurement
  2. . Record BP readings in their diary
  Hypertensive patient on usual care: Patient do home BP monitoring Record the Home BP monitoring in their diary
- Total: Total of all reporting groups
Arm/Group | Smart Phone Based Telemonitoring of HBP | Hypertensive Patients on Usual Care | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (8.7) | 59.4 (8.9) | 58.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 51 | 51 | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 105 | 105 | 210
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 105 | 105 | 210

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Doing Home BP Monitoring
Description: Percentage of subjects doing home BP monitoring with at least BP recordings of three or more times/week
Time Frame: Baseline, 3rd month, 6th month
Measure: Number; unit: percentage of subjects doing HBPM
Groups:
- Hypertensive Patients on Enhanced Usual Care: Hypertensive patients on usual care
  1. . Patients to do HBP measurement
  2. . Record BP readings in their diary
  Hypertensive patient on usual care: Patient do home BP monitoring Record the Home BP monitoring in their diary
Arm/Group | Smart Phone Based Telemonitoring of HBP | Hypertensive Patients on Enhanced Usual Care
Number analyzed (Participants) | 105 | 105
percentage of subjects doing HBPM
  baseline | 54 | 46
  3rd month | 68 | 64
  6th month | 67 | 62
Statistical Analysis 1: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; comparison of the percentage of patients doing HBPM between intervention and control group at baseline; Test type: Superiority or Other; p = 0.27, Chi-squared
Statistical Analysis 2: Comparison: Smart Phone Based Telemonitoring of HBP; Comparison of percentage of subjects doing HBPM at 3rd month from baseline within intervention group; Test type: Superiority or Other; p = .020, McNemar
Statistical Analysis 3: Comparison: Smart Phone Based Telemonitoring of HBP; comparison in percentage of patients doing Home BP monitoring at 6th month from baseline within intervention group; Test type: Superiority or Other; p = .060, McNemar
Statistical Analysis 4: Comparison: Hypertensive Patients on Enhanced Usual Care; Change in the proportion of patients doing HBPM at 3 months from baseline within the control group; Test type: Superiority or Other; p = .002, McNemar
Statistical Analysis 5: Comparison: Hypertensive Patients on Enhanced Usual Care; Change in proportion of patients doing HBPM at 6 months from baseline within control group; Test type: Superiority or Other; p = .009, McNemar

2. Primary Outcome: Change in Mean Clinic Systolic and Diastolic Blood Pressure CSBP and CDBP Readings at 3 and 6 Months From Baseline
Description: At baseline and follow-up visits, research assistants who are blinded to allocation outcomes will meaure blood pressure after 15 minutes rest with validated electronic automated sphygmanometer ( ) . Four blood pressure readings taken at 1 minute interval will done for each subject and the mean of the second and third reading would be used for the primary outcome ,
Time Frame: baseline, 3rd month and 6 month
Population: Intention to treat analysis was used and the last known data were carried forward to replace missing values for drop-outs.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Smart Phone Based Telemonitoring of HBP | Hypertensive Patients on Enhanced Usual Care
Number analyzed (Participants) | 105 | 105
mmHg
  baseline mCSBP in mmHg | 129.96 (11.86) | 130.40 (14.74)
  baseline mCDBPin mmHg | 81.19 (8.49) | 81.41 (10.12)
  change mCSBPat 3 months | -2.22 (15.3) | -3.28 (13.9)
  change in mCDBP at 3 months | -2.42 (7.4) | -0.82 (8.8)
  change mCSBP 6 months from baseline | -1.10 (13.1) | -2.82 (14.4)
  change mCDBPat 6 months from baseline | -1.35 (6.2) | -1.52 (8.7)
Statistical Analysis 1: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; Comparison of baseline mean clinic systolic BP mCSBP readings between control and intervention; Test type: Superiority or Other; p = 0.813, t-test, 2 sided
Statistical Analysis 2: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; Comparison of baseline mean clinic diastolic BP mCDBP readings between control and intervention; Test type: Superiority or Other; p = 0.865, t-test, 2 sided
Statistical Analysis 3: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; Comparison of difference of mean clinic systolic BP readings mCSBP between control and intervention at 3 months from baseline; Test type: Superiority or Other; p = 0.476, t-test, 2 sided
Statistical Analysis 4: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; Comparison of difference of mean clinic diastolic BP mCDBP readings between control and intervention at 3 months from baseline; Test type: Superiority or Other; p = 0.14, t-test, 2 sided
Statistical Analysis 5: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; Comparison of difference of mean clinic systolic BP readings mCSBP between control and intervention at 6 months from baseline; Test type: Superiority or Other; p = 0.495, t-test, 2 sided
Statistical Analysis 6: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; Comparison of difference in mean clinic diastolic BP readings mCDBP between control and intervention at 6 months from baseline; Test type: Superiority or Other; p = 0.967, t-test, 2 sided

3. Secondary Outcome: Self-efficacy for Managing Chronic Disease: 6 Items Scale (SEMCD-6 Items) Comparing Both Groups at 3 and 6 Months Post-intervention
Description: This is a 6-items scale for measuring confidence of patients in self management of their chronic disease. Each item has a likert scale from 1 to 10 with 10 as most confident. Higher score indicating higher self-efficacy
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smart Phone Based Telemonitoring of HBP + Enhanced Usual Care | Hypertensive Patients on Enahnced Usual Care
Number analyzed (Participants) | 105 | 105
units on a scale
  baseline SEMCD between groups | 37.72 (11.59) | 38.10 (11.85)
  3 months SEMCD from Baseline between groups | 39.99 (10.07) | 38.96 (10.43)
  6 months SEMCD from baseline between groups | 38.75 (10.92) | 37.74 (11.36)
Statistical Analysis 1: Comparison: Smart Phone Based Telemonitoring of HBP + Enhanced Usual Care vs Hypertensive Patients on Enahnced Usual Care; Comparison of baselline SEMCD between telemonitoring group and enhanced usual care; Test type: Superiority or Other; p = 0.819, t-test, 2 sided
Statistical Analysis 2: Comparison: Smart Phone Based Telemonitoring of HBP + Enhanced Usual Care vs Hypertensive Patients on Enahnced Usual Care; Comparison of SEMCD at 3 months between telemonitoring group and enhanced usual care; Test type: Superiority or Other; p = 0.512, t-test, 2 sided
Statistical Analysis 3: Comparison: Smart Phone Based Telemonitoring of HBP + Enhanced Usual Care vs Hypertensive Patients on Enahnced Usual Care; Comparison of SEMCD at 6 months between telemonitoring group and enhanced usual care group; Test type: Superiority or Other; p = 0.325, t-test, 2 sided

4. Primary Outcome: Comparison of Mean Home Systolic and Diastolic Blood Pressure mHSBP and mHDBP Readings Between Intervention and Control Grp at Baseline
Description: At baseline and follow-up visits, research assistants will collect the HSBP and HSBP readings of both groups at baseline, 3rd and 6th month FU. Regular home BP measurement is taken as the average of at least 3 or more BP measurement readings per week. The research assistant are not blinded and will collect the average of paper SBP and DBP measurement recordings ( if done) of the control group at baseline,at 3rd month and 6th month. The research assistant are not blinded and will collect the average of smartphone based SBP and DBP measurement recordings ( if done) and sent to the data center of the intervention group at baseline,at 3rd month and 6th month.
Time Frame: baseline
Population: The mean average of the HSBP and HDBP of both groups who have taken and recorded their blood pressure readings at least 3x or more per week are collected
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Smart Phone Based Telemonitoring of HBP | Hypertensive Patients on Enhanced Usual Care
Number analyzed (Participants) | 93 | 79
mmHg
  baseline HSBP in mmHg | 127.17 (11.08) | 128.35 (13.53)
  baseline HDBPin mmHg | 77.16 (8.13) | 77.32 (8.31)
Statistical Analysis 1: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; comparison of baseline mHSBP in mmHg between Telemonitoring and Enhanced Usual Care groups; Test type: Superiority or Other; p = 0.532, t-test, 2 sided
Statistical Analysis 2: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; comparison of baseline mHDBP in mmHg between Telemonitoring and Enhanced Usual Care groups; Test type: Superiority or Other; p = 0.902, t-test, 2 sided

5. Primary Outcome: Comparison of Mean Home Systolic and Diastolic Blood Pressure mHSBP and mHDBP Readings at 3 Months Between Smart Phone Based Telemonitoring Group and Control Group on Enhanced Usual Care
Description: as for outcome 4
Time Frame: 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Smart Phone Based Telemonitoring of HBP | Hypertensive Patients on Enhanced Usual Care
Number analyzed (Participants) | 104 | 97
mmHg
  3 months HSBP in mmHg | 121.50 (11.17) | 124.37 (10)
  3 months HDBPin mmHg | 73.93 (7.24) | 74.97 (7.91)
Statistical Analysis 1: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; comparison of mHSBP at 3 months between smartphone based telemonitoring group and control group on enhanced usual care; Test type: Superiority or Other; p = 0.138, t-test, 2 sided
Statistical Analysis 2: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; comparison of mHDBP in mmHg between Telemonitoring and Enhanced Usual Care groups at 3 months; Test type: Superiority or Other; p = 0.204, t-test, 2 sided

6. Primary Outcome: Comparison Between Mean Home Systolic and Diastolic Blood Pressure HSBP and HDBP Readings at 6 Months Between the Smartphone Based Telemonitoring Group and Control Group on Enhanced Usual Care
Description: as for outcome 4
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Smart Phone Based Telemonitoring of HBP | Hypertensive Patients on Enhanced Usual Care
Number analyzed (Participants) | 102 | 94
mmHg
  mHSBP in mmHg at 6 months between groups | 122.63 (11.1) | 124.95 (11.25)
  mHDBPin mmHg at 6 months between groups | 74.15 (8.23) | 75.87 (7.59)
Statistical Analysis 1: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; comparison of mHSBP in mmHg between Telemonitoring groups and Enhanced Usual Care groups at 6 months; Test type: Superiority or Other; p = 0.199, t-test, 2 sided
Statistical Analysis 2: Comparison: Smart Phone Based Telemonitoring of HBP vs Hypertensive Patients on Enhanced Usual Care; comparison of mHDBP in mmHg at 6 months between Telemonitoring and Enhanced Usual Care groups; Test type: Superiority or Other; p = 0.204, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Smart Phone Based Telemonitoring of HBP: 1. . Patients do HBP monitoring
  2. . record their BP readings into the smart phone with downloaded application.
  Smart phone telemonitoring HBP + enhanced usual care: Smart phone telemonitoring home Blood pressure (HBP) Patients input their HBP readings to their smart phone which is sent to the data center regulary
- Enhanced Usual Care: 1. . Patients to do HBP measurement
  2. . Record BP readings in their diary
  Enhanced usual care: Encouraged to do HBP measurement and record BP readings in paper diary
Arm/Group | Smart Phone Based Telemonitoring of HBP | Enhanced Usual Care
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 0/105 | 0/105

LIMITATIONS AND CAVEATS:
The baseline mean Clinic SBP and DBP as well as the baseline mean home SBP and DBP of both the control and intervention group were already within the optimal range.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No